CLINICAL TRIAL: NCT06797128
Title: Comparison of Bicep Tendon Migration Between Two Techniques for Open Subpectoral Biceps Tenodesis
Brief Title: Comparison of Two Surgical Techniques for Open Subpectoral Biceps Tenodesis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Michael T. Freehill, Associate Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 77635
Record Dates: First submitted 2025-01-21; First posted 2025-01-28 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Bicep Tenodesis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- One Anchor (Experimental): Participant will receive one standard anchor during standard biceps tenodesis procedure
  Interventions: Procedure: One Anchor
- Two Mini Anchors (Experimental): Participant will receive two mini anchors during standard biceps tenodesis procedure
  Interventions: Procedure: Two Mini Anchors

INTERVENTIONS:
Procedure: One Anchor — Participant will receive one standard anchor
  Arms: One Anchor
Procedure: Two Mini Anchors — Participant will receive two mini anchors
  Arms: Two Mini Anchors

SUMMARY:
Participants who are indicated for an open biceps tenodesis procedure will be recruited to join the study. The participant will undergo the standard biceps tenodesis procedure using either one standard anchor or two mini anchors by the study staff surgeon. Both techniques are safe and considered standard of care. The participant will be randomized to either group. After the biceps are secured in the standard fashion, a sterile radiolucent bead will be applied to the tendon. The participant will undergo xray imaging in the post-anesthesia care unit to determine a baseline measurement of the location of the radiolucent bead. The participant will then undergo further xray imaging at their 2 week and 6 month-up visits.

DETAILED DESCRIPTION:
Participants who are indicated for an open biceps tenodesis procedure will be recruited to join the study. The participant will undergo the standard biceps tenodesis procedure using either one standard anchor or two mini anchors by the study staff surgeon. Both techniques are safe and considered standard of care. The participant will be randomized to either group. After the biceps are secured in the standard fashion, a sterile radiolucent bead will be applied to the tendon. This will allow for measurements to be made on xray imaging in the post-operative period. The placement of the clip is the only experimental portion of the procedure. The participant will undergo xray imaging in the post-anesthesia care unit to determine a baseline measurement of the location of the radiolucent bead. The participant will then undergo further xray imaging at their 2 week and 6 month-up visits. These visits are standard visits for the participant who undergo this procedure.

ELIGIBILITY:
Inclusion Criteria:

* Participant age 18 and above who would otherwise indicated for biceps tenodesis due to biceps tendinopathy with or without associated rotator cuff pathology

Exclusion Criteria:

* Participant under the age of 18 will be excluded from the study as there is no indication to perform this procedure in children.
* Any participant who had previous surgery or injury to their biceps or biceps tendon will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Sterile radiolucent bead location distance | Baseline, 2-weeks, 6-months
  Sterile radiolucent bead location will be measured during all 3 xrays. Comparison of these measurements will be between the two groups.

SECONDARY OUTCOMES:
Participant Reported Outcome VAS | 2-weeks, 6-months
  Change in Visual Analog Scale (VAS); minimum 0, maximum 10, higher score is a worse outcome
Participant Reported Outcome Constant | 2-weeks, 6-months
  Constant Score; minimum 0, maximum 100, higher score is a better outcome
Participant Reported Outcome ASES | 2-weeks, 6-months
  American Shoulder Elbow Score (ASES); minimum 0, maximum 100, higher score is a better outcome
Participant Reported Outcome SSV | 2-weeks, 6-months
  Subjective Shoulder Value (SSV); minimum 0, maximum 100, higher score is a better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Michael Freehill, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No